CLINICAL TRIAL: NCT06968416
Title: 12-Week Efficacy Clinical Study of Serum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C23005030
Record Dates: First submitted 2025-04-21; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Anti-aging; Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group Serum (Other): 65 female adult subjects will be enrolled in the study, recruited according to inclusion and non-inclusion criteria listed below, at least 40 subjects should complete the clinical evaluation and image capture, 60 subjects should complete consumer questionnaire.
  Interventions: Other: Standard cleanser，standard moisturizer，standard sunscreen，Investigational serum

INTERVENTIONS:
Other: Standard cleanser，standard moisturizer，standard sunscreen，Investigational serum — Products Application and Usage Instruction
  1. Mode of application: T-3W ~ T0
     Frequency:
     AM: Standard cleanser + standard moisturizer + standard sunscreen PM: Standard cleanser + standard moisturizer Caution: No any other skincare or facial make up products are used except provide products
  2. Mode of application: T0 ~ T12W
  Frequency:
  AM: Standard cleanser + Investigational serum (face and eye) [FLA #774715 21] + standard moisturizer + standard sunscreen PM: Standard cleanser + Investigational serum (face and eye) [FLA #774715 21] + standard moisturizer
  Caution: No any other skincare or facial make up products are used except provide products
  Usage Instruction： Use serum [FLA #774715 21] 8-10 drops (0.3ml) on cleansed face and eye skin 2 times a day (AM & PM).

SUMMARY:
65 female adult subjects will be enrolled in the study, recruited according to inclusion and non-inclusion criteria listed above. At least 40 subjects should complete the clinical evaluation and 60 subjects should complete consumer questionnaire in this 15-week study (wash-out phase for 3 weeks and treatment phase for 12 weeks). Subjects will need to refrain from using any product other than the provided test products on whole face including eye area during the 3-week wash-out phase and 12-week study treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged from 25-55 years old.
2. All skin types, including 50% sensitive skin.
3. Regular users of serum with anti-aging need.
4. Self-claim concerns of skin quality problem (radiance, smoothness, pore) and aging problems (fine lines, wrinkles, elasticity).
5. Presenting with corresponding severity for the attribute evaluated by Dermatologist： Crows' feet wrinkle (Loreal atlas, 2≤grade≤5) Underneath Eye Wrinkle (Loreal atlas, 2≤grade≤5) Inter Ocular Wrinkles (Loreal atlas, 1<grade≤4) Glabellar wrinkles (Loreal atlas, 1<grade≤4) Nasolabial fold (Loreal atlas, 2≤grade≤4) Forehead wrinkle (Loreal atlas, 2≤grade≤5) Fine lines on the forehead (Loreal atlas, 1<grade≤4) Cheek folds (Loreal atlas, 2≤grade≤5) Wrinkles of the corner of the lips (Loreal atlas, 1<grade≤4)
6. Clinical grading of skin pores, skin radiance and skin smoothness: 4≤grade≤6 evaluated by dermatologist.
7. No disagreement of dermatologist because of other reasons that exclude the participation of the subject.
8. In general good health at the time of the study.
9. Willing and able to participate as evidenced by signing of informed consent and photo release form.
10. Must be willing to comply with all study protocol requirements (pay attention to: only use the provided product during the study, not take topical or oral treatment like retinol, hormone, anti-oxidant health-care products which may impact the efficacy of study).

Exclusion Criteria:

1. Pregnant or breast-feeding woman or woman planning pregnancy during the study.
2. Subject deprived of rights by a court or administrative order.
3. Major subject to a guardianship order.
4. Subject residing in a health or social care establishment.
5. Patient in an emergency setting.
6. Subject with a skin disease in the test areas (particularly e.g., acne, rosacea, eczema).
7. Subject presenting a stable or progressive serious disease (per investigator's assessment).
8. Immuno-compromised subject.
9. Subject with history of allergy to cosmetic or personal care products or ingredients.
10. Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).
11. Subjects regularly practicing aquatic or nautical sports.
12. Subjects regularly attending a sauna.
13. Subject with cardiovascular or circulatory history.
14. Subject with a history of skin cancer or malignant melanoma.
15. Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Time effect of skin smoothness (Visual) | Compare to baseline，Time point immediate , Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of skin radiance (Visual) | Compare to baseline，Time point immediate , Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of skin pore (Visual) | Compare to baseline，Time point immediate , Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of skin elasticity (Tactile) | Compare to baseline，Time point immediate , Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of skin firmness (Visual) | Compare to baseline，Time point immediate , Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of forehead wrinkles | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of fine lines on the forehead | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of glabellar wrinkles | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of inter-ocular wrinkles | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of crow's feet wrinkles | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of underneath eye wrinkles | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of cheek folds | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of nasolabial fold | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of wrinkles of the corner of the lips | Compare to baseline，Time point at 1Week , Time point at 2Week, Time point at 4Week, Time point at 8Week and Time point at 12Week.

SECONDARY OUTCOMES:
Time effect of count number of forehead wrinkles by Primos | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of total length of forehead wrinkles by Primos | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of area of forehead wrinkles by Primos | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of count number of crow's feet wrinkles by Primos | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of total length of crow's feet wrinkles by Primos | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of area of crow's feet wrinkles by Primos | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of thickness of dermis by UC22 | Compare to baseline，Time point at 8Week and Time point at 12Week.
Time effect of thickness of epidermis by UC22 | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.
Time effect of thickness of epidermis and dermis by UC22 | Compare to baseline，Time point at 4Week, Time point at 8Week and Time point at 12Week.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Xu, Master, Principal Investigator — Shanghai China-norm Quality Technical Service Co., Ltd.
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon PRS registration completion.
  Timeline:
  Months 1-2: Data de-identification, metadata preparation, and platform integration.
  Month 3: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn